CLINICAL TRIAL: NCT04798274
Title: Role of GABAergic Transmission in Auditory Processing in Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 200159; 20-M-0159
Record Dates: First submitted 2021-03-12; First posted 2021-03-15 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11-28

CONDITIONS: Autism Spectrum Disorder
Keywords: GABA; Language; ASD; MEG; MRS
MeSH Terms: conditions — Autism Spectrum Disorder; Language

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active cTBS (Experimental): This intervention involves active repetitive magnetic stimulation. The coil emits a magnetic field
  Interventions: Device: Continuous Theta Burst Stimulation
- Sham cTBS (Sham Comparator): This intervention involves sham (placebo) repetitive transcranial magnetic stimulation. The coil is blinded, but does not emit any magnetic field
  Interventions: Device: Continuous Theta Burst Stimulation

INTERVENTIONS:
Device: Continuous Theta Burst Stimulation — Continuous theta burst stimulation (cTBS) will be applied using a MagPro X100 (MagVenture, Inc. Alpharetta, GA). The cTBS protocol consists of bursts of three pulses of 50 Hz stimulation repeated at 200 ms intervals (5 times per second) for 40 seconds (for a total of 600 pulses). Stimulation will be applied at an intensity of 80% of active motor threshold (AMT). Brainsight (Rogue Research) frameless neuronavigation system will be used to target the specific structural MRI-defined region of stimulation.

SUMMARY:
Background:

Autism spectrum disorder (ASD) is a complex neurodevelopmental syndrome. Researchers think brain development may be controlled by gamma-aminobutyric acid (GABA). They want to learn how abnormalities in the GABA system may contribute to ASD.

Objective:

To see if repetitive transcranial magnetic stimulation (rTMS) creates short-term changes in how different parts of the brain communicate.

Eligibility:

Right-handed people ages 11-17 with ASD, and healthy volunteers ages 18-25.

Design:

Participants will be screened with:

Medical history

Physical exam

Medicine review

Neurological exam

Psychological tests and rating scales

Forms and surveys.

Participants will have a hearing test and ear exam.

Participants will have magnetic resonance imaging (MRI) of the brain. They will lie on a table that moves in and out of the MRI scanner. They may look at a screen while in the scanner. A coil will be placed over their head.

Participants will have magnetic resonance spectroscopy. It takes pictures of chemicals in the brain using the MRI scanner.

Participants will have magnetoencephalography. They will sit in a chair. A helmet with magnetic field sensors will be placed on their head.

Participants will have TMS. A wire coil will be held on their scalp. A brief electrical current will pass through the coil.

Participants will have electromyography. Sticky pad electrodes will be placed on the skin during TMS. The electrical activity of their muscles will be measured.

Participants will have rTMS. It uses short bursts of magnetic pulses to affect brain activity.

ASD participants may have visits scheduled as often as 1 time a week or as far apart as 2 months based on the participants or study team's availability. Healthy volunteers will have 3 visits over 3-4 weeks....

DETAILED DESCRIPTION:
Study Description:

This will be a within-subject, controlled, proof-of-mechanism study.

Objectives:

The study aims to evaluate the relationship between local GABA concentration, structural and functional network connectivity and MEG measures of auditory and language processing in adolescents with ASD and the acute impact of a single session of continuous theta burst stimulation over left posterior superior temporal cortex (pSTC) on these measures. We hypothesize that GABA concentrations, DWI measures of tissue microstructure and fcMRI obtained BOLD correlations within the language network will significantly contribute to the prediction model for MEG indices of auditory and language processing. Participation in the study involves about seven study visits. Some of the visits may be split up to shorten the length of session and limit fatigue. Visits may be scheduled as frequent as about once a week or as far apart as two months per the patient or study team's availability. All visits must be completed within six months of the date of enrollment.

Primary Objective: The overall goal of the current study is to 1) Characterize the relationship between an individual's baseline local cortical GABA concentration, DWI measures of auditory and language network tissue microstructure, and fcMRI indices of local and long-range network functional connectivity (predictor variables) and MEG indices of auditory and language processing (dependent variables).

Secondary Objectives: 2) Evaluate the impact of a single session of cTBS over the left pSTC on these MRS and MEG indices in adolescents (age 11-17) with ASD.

Exploratory Objective: 3) Characterize the relationship between the neuroimaging and electrophysiological indices obtained in this study and baseline behavioral symptom presentation.

Endpoints:

Primary Endpoints:

1. MEG: Evoked fields and Spectral Power
2. MRS: GABA+/Cr concentrations in the left pSTC
3. DWI: Diffusion derived parameters in the auditory radiations and arcuate fasciculus.
4. fcMRI: BOLD correlations across pre-defined ROIs.

Secondary Endpoints:

a. MEG: Inter-trial gamma-band coherence (ITC) and resting state alpha to gamma phase-amplitude coupling.

Exploratory Endpoints:

a. SRS-2, CELF-5, EVT-3, PPVT-5, ADOS-2 (if available), ADI-R, VABS-III, WASI-II, CBCL, EDI.

ELIGIBILITY:
* INCLUSION CRITERIA:

Pilot Phase

Inclusion criteria

* Ability to provide informed consent
* Age: 18-25 years
* Must meet the definition of "Healthy Control" having completed the screening assessment under protocol 01-M-0254, "The Evaluation of Patients with Mood and Anxiety Disorders and Healthy Volunteers" or under protocol 17-M-0181, "Recruitment and Characterization of Research Volunteers for NIMH Intramural Studies".

Main Study Phase

Inclusion criteria

* Ability to provide informed assent and parent consent (Parents of children enrolling on the study do not need to be able to speak English. A consent form is available in English or Spanish for parents of children who enroll.)
* Age: 11-17 years
* Community Diagnosis of ASD based on DSM-IV or DSM-5 criteria (reviewed by a member of the Neurodevelopmental and Behavioral Phenotyping Service)
* Wechsler Abbreviated Scale of Intelligence, Second Edition (WASI-II). WASI-II will be used as a measure of intellectual function. Children will be included when FSIQ > 70.
* Right-handed: to reduce heterogeneity.
* Hearing: Normal hearing in order to complete the behavioural assessments.

EXCLUSION CRITERIA:

Participants will be screened to exclude individuals with co-occurring neurological or medical conditions that might confound the results, as well as to exclude subjects in whom MRI or rTMS might result in increased risk of side effects or complications. This accounts for the majority of the exclusion criteria listed:

Exclusion criteria

Participants will be screened to exclude individuals with neurological, psychological/behavioral or medical conditions, as well as to exclude subjects in whom MRI or rTMS might result in increased risk of side effects or complications. This accounts for the majority of the exclusion criteria listed:

Pilot Phase

* Non-English Speakers
* Known Neurological Disorder
* Known Psychiatric Disorder
* Known genetic disorder (e.g., NF1, tuberous sclerosis), acquired neurologic disease (e.g. stroke, tumour), cerebral palsy, intracranial pathology or significant dysmorphology;
* History of fainting spells of unknown or undetermined etiology that might constitute seizures;
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy;
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.);
* Past or Current History of Tinnitus
* Any implant, prosthesis or other permanent alteration of the body that, in the opinion of the investigator, would be unsafe with MRI or TMS or that would produce an artifact that would compromise the integrity of data;
* Signs of increased intracranial pressure;
* Intracranial lesion (including incidental finding on MRI) that, in the opinion of the investigator, would be unsafe with MRI or TMS or that would produce an artifact that would compromise the integrity of data;
* History of any head trauma within 6 months of screening, or beyond 6 months prior to screening, history of head trauma with evidence of traumatic abnormality appearing on a brain scan, or with loss of consciousness >5 minutes, or with other sequelae, excluding headache, lasting > 24 hours.
* Pregnancy;
* Participants who have received rTMS less than 7 days prior to enrollment;
* Individuals currently taking GABAergic medications or any other medication that, in the opinion of the investigator, significantly lowers seizure threshold;
* Individuals for whom it is not safe or appropriate to remain on a stable pharmacotherapy (for nonexclusionary medications) for six weeks prior to and over the course of their participation in the study;
* A current NIMH employee or staff or their immediate family member.

Main Study Phase

* Non-English Speakers
* Known genetic disorder that is either associated with the ASD diagnosis or that in the opinion of the investigator may increase the risk to the participant or compromise the integrity of the data;
* Acquired neurologic disease (e.g. stroke, tumour), cerebral palsy, intracranial pathology or significant dysmorphology;
* History of fainting spells of unknown or undetermined etiology that might constitute seizures;
* History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy;
* Any progressive (e.g., neurodegenerative) neurological disorder;
* Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.);
* Past or Current history of clinically significant tinnitus as determined by an audiologist or other-licensed clinician.
* Any implant, prosthesis or other permanent alteration of the body that, in the opinion of the investigator, would be unsafe with MRI or TMS or that would produce an artifact that would compromise the integrity of data;
* Signs of increased intracranial pressure;
* Intracranial lesion (including incidental finding on MRI) that, in the opinion of the investigator, would be unsafe with MRI or TMS or that would produce an artifact that would compromise the integrity of data;
* History of any head trauma within 6 months of screening, or beyond 6 months prior to screening, history of head trauma with evidence of traumatic abnormality appearing on a brain scan, or with loss of consciousness >5 minutes, or with other sequelae, excluding headache, lasting > 24 hours.
* Pregnancy;
* Participants who have received prior rTMS;
* Active or History of psychosis, bipolar disorder, active severe substance use disorders (within the last month), have active suicidal intent or plan as detected on screening instruments or in the investigator team's opinion is likely to attempt suicide within 6 months;
* Individuals currently taking GABAergic medications or any other medication or medication change that, in the opinion of the investigator, significantly lowers seizure threshold;
* Past or present medical or neurological condition, disease, disorder, genetic finding, or injury that, in the opinion of the Investigator, may significantly increase the potential risks of study participation, reduce or compromise a subject's ability to fully comply with all study requirements for the duration of the study or may compromise the integrity of the data.

Ages: 11 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 106 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
MRS | immediately pre and post rTMS
  GABA+/Cr concentrations in the left pSTC
MEG | immediately pre and post rTMS
  Evoked fields and Spectral Power
fcMRI | immediately pre and post rTMS
  BOLD correlations across pre-defined ROIs.
DTI | immediately pre and post rTMS
  Diffusion tensor derived parameters in the auditory radiations and arcuate fasciculus.

SECONDARY OUTCOMES:
Neuropsychological Assessments | Baseline
  SRS-2, CELF-5, EVT, PPVT, ADOS-2, ADI-R, VABS-III, WASI-II.
MEG | immediately pre and post rTMS
  Inter-trial gamma-band coherence (ITC) and resting state alpha to gamma phase-amplitude coupling.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Pine, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-M-0159.html